CLINICAL TRIAL: NCT04431882
Title: The Role of Optic Nerve Sheath Fenestration in Leukemic Patients Having Increased Intracranial Pressure
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Fahmy Doheim, Dr., Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304628
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Leukemic Patients With Increased Intracranial Pressure; Optic Nerve Sheath Fenestration

STUDY DESIGN:
Intervention Model Description: A single arm clinical trial for patients presenting with severe sight threatening papilledema due increased intracranial pressure following leukemia treatment meeting the criteria of idiopathic intracranial hypertension not responding to maximal medical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- optic nerve sheath fenestration (Experimental): Leukemic patients mainly those suffering from acute lymphoblastic leukemia.
  Interventions: Procedure: optic nerve sheath fenestration

INTERVENTIONS:
Procedure: optic nerve sheath fenestration — A standard medial transconjunctival orbitotomy was performed in all cases under general anesthesia. The medial rectus muscle was disinserted and reflected nasally with 6-0 synthetic polyester suture in typical fashion for eye muscle surgery. A traction suture was then placed through the insertion stump of the medial rectus in a baseball stitch fashion to facilitate abduction of the globe. The pupil was monitored at all times. A custom- made cupped orbital retractor was inserted along the medial scleral wall and used to retract the orbital fat and allow visualization of the optic nerve sheath. Retraction and globe abduction were relaxed if any changes in pupil size were noted. When adequate visualization was achieved, multiple dural sheath fenestrations approximately 3 mm in length. Expulsion of cerebrospinal fluid was invariably observed with the initial incision into the dural sheath.

SUMMARY:
Optic nerve sheath fenestration (ONSF) first described by De Wecker in 1872 for the treatment of neuroretinitis. Since then, optic nerve sheath fenestration has become well established procedure for treatment of papilledema in medically uncontrolled patients of idiopathic intracranial hypertension.

DETAILED DESCRIPTION:
Optic nerve sheath fenestration (ONSF) first described by De Wecker in 1872 for the treatment of neuroretinitis. Since then optic nerve sheath fenestration has become well established procedure for treatment of papilledema in medically uncontrolled patients of idiopathic intracranial hypertension. Indications for ONSF in cancer patients are not well established, but a few case reports have shown success of ONSF in patients with perineural metastasis of breast cancer, increased intracranial pressure with papilledema due to a brain tumor, leukemia and optic nerve sheath meningioma. This study is conducted to establish the role of optic nerve sheath Fenestration in leukemic patients mainly those suffering from acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of progressive visual loss and papilledema did not improve despite the maximal medical therapy prescribed.
* Informed written consent was obtained from the parents/care providers of the study participants.

Exclusion Criteria:

* Can not get the informed consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity using LOGMAR | Three months
  Visual acuity using LOGMAR
Papilledema grading using frisén scale | Three months
  Papilledema grading using frisén scale

SECONDARY OUTCOMES:
Visual acuity using LOGMAR | 2 weeks
  Visual acuity using LOGMAR
Papilledema grading using frisén scale | 2 weeks
  Papilledema grading using frisén scale

CONTACTS AND LOCATIONS:
Overall Officials: Mai ElBahwash, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data shared upon request from the corresponding author